CLINICAL TRIAL: NCT05123300
Title: PRISMA-PET - Primary Staging of Prostate Cancer: A Randomized Controlled Trial Comparing 18F-PSMA-1007 PET/CT to Conventional Imaging
Brief Title: PRISMA-PET - Primary Staging of Prostate Cancer With PSMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to change of EAU guidelines, where PSMA-PET/CT is now recommended for primary staging of prostate cancer. We do not believe we ethically could continue this protocol, when the new examination, that was our intervention, is now the recommended.
Sponsor: Odense University Hospital (Other)
Collaborators: Sygehus Lillebaelt (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Karen Middelbo Buch-Olsen, physician, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020110469
Record Dates: First submitted 2021-08-31; First posted 2021-11-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Primary staging; PSMA-PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Included patients will be randomized 1:1 into a control group (A) and an interventional group (B). Block randomization will be stratified by high-/intermediate-/low-risk PCa patients. Bone Scan has been substituted with NaF-PET/CT in clinical routine at participating departments, and will as well in this study.
  Primary staging in each group will be performed as follows:
  * Group A: CE-CT and NaF-PET/CT (conventional imaging)
  * Group B: 18F-PSMA-1007 PET/CT (interventional imaging) In group B, a sufficient number of patients will have conventional imaging performed (an added NaF-PET/CT), which will be blinded and used for diagnostic accuracy measures. A subset of patients with risk of extracapsular extension planned for radical prostatectomy in group B will also have an 18F-PSMA-PET/MRi-scan performed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A) Conventional Imaging (No Intervention): Conventional Imaging with NaF (sodium fluoride)-PET/CT used for staging
- B) Interventional Imaging (Experimental): Staging with the interventional18F-PSMA-1007 PET/CT.
  Interventions: Diagnostic Test: 18F-PSMA-1007

INTERVENTIONS:
Diagnostic Test: 18F-PSMA-1007 — 18F-PSMA-1007 is a tracer for a PET/CT. Prostate cancer often has marked uptake of PSMA, hence PSMA-PET/CT is in the guidelines in the European Union for detecting relapse. But we will use it for staging primary prostate cancer.
  Arms: B) Interventional Imaging

SUMMARY:
Early and correct diagnostic staging is paramount to keep patients with newly diagnosed prostate cancer in the correct treatment tract to avoid under- and overdiagnosis in prostate cancer staging. With accurate staging, the investigators aim to save patients from side effects of insufficient or too extensive treatment. The investigators hypothesize that precise staging will lead to optimized individualized treatment and subsequently to prolonged survival and increased quality of life.

Prostate cancer is a very heterogeneous disease varying from indolent tumors to aggressive cancer types. About one-fifth of patients with newly detected high- or intermediate-risk prostate cancer present with bone metastases and their 3-years survival is less than 50%. Precise staging is required for planning relevant treatment that has the potential to increase survival.

The prostate-specific membrane antigen (PSMA) is overexpressed in prostate cancer cells and can serve as a target for precise diagnosis and staging. PSMA-positron emission tomography/computed tomography (PET/CT) has shown to be more accurate than traditional imaging, but there is a need for prospective trials analyzing the impact of primary staging with PSMA-PET/CT on treatment planning and patient benefit.

In a prospective multicenter study, the investigators plan to include 448 patients and randomize 1:1 to either traditional imaging or PSMA-PET/CT. The investigators aim to analyze whether PSMA-PET/CT increases progression-free survival and quality of life. Further, the investigators aim to validate the accuracy of primary staging with PSMA-PET/CT compared with conventional imaging.

DETAILED DESCRIPTION:
Introduction

The proposed project shall reveal whether primary staging with up-to-date imaging benefits prostate cancer (PCa) patients in terms of yielding prolonged progression-free survival and increased quality of life (QoL).

The study is planned in a collaborative effort between five centers in the Region of Southern Denmark and the Central Denmark Region. The Department of Nuclear Medicine at Odense University Hospital is the hosting department.

A prospective multicenter randomized design is planned. We expect to include 448 patients with newly diagnosed PCa of high or intermediate risk. Eligible patients will be randomized 1:1 into an interventional arm using PSMA-PET/CT and a control arm using conventional imaging. In a relevant subgroup, the investigators will also analyze the added value of performing PSMA-PET/magnetic resonance imaging (MRi).

The investigators hypothesize that PSMA-PET/CT will lead to prolonged progression-free survival and increased quality of life when used for staging patients with intermediate and high-risk primary prostate cancer.

Background

Prostate Cancer (PCa) is the most frequent cancer form in men, and approximately 4,500 new cases are reported each year in Denmark. The course of disease ranges from slow-growing tumors localized to the prostate gland itself to aggressive, rapidly disseminating variants. Aggressive variants of the disease can be disseminated initially, e.g. to lymph nodes or bone. The overall 5-year survival is as high as 87% for the broad group of PCa patients, but for patients diagnosed with bone metastases initially, the prognosis is poor with a 3-year survival of 62%. It is currently widely debated whether these patients should be managed using systemic therapies or aggressive local and metastases-directed therapies. Early and correct staging is paramount to get this closer, hence aiming to avoid under- and overtreatment.

Curatively intended surgery or radiation treatment is the initial intervention for patients with localized disease, while androgen deprivation or chemotherapy is recommended for patients with metastatic disease in current guidelines. As regards the primary staging of PCa, the guidelines recommend traditional imaging, including bone scan (BS) and contrast enhanced CT (CECT), and these are rather inaccurate. BS reflects bone metabolism and has a reported sensitivity as well as specificity of 80%. An emerging modality also reflecting bone metabolism is the 18Fluoride(18F)-sodium fluoride(NaF)-PET/CT, but this method has not proven any added value compared with BS.

The transmembrane protein, PSMA, is expressed in abundance on the surface of prostate cancer cells, and this has become a unique target for accurate diagnosis and is already implemented for imaging in recurrent PCa. The PSMA ligands are labeled with positron-emitting isotopes such as 18F and 68Gallium(68Ga) for imaging. The 18F isotope is advantageous regarding availability and production, and the 18F-labeled ligand, PSMA-1007, is only sparsely excreted in the urinary tract, making diagnostics in the pelvic region favorable.

Diagnostic accuracy studies performed in the primary PCa setting have been published recently. A retrospective Danish study of 68Ga-PSMA-PET/CT in the so-far largest cohort of 691 patients with newly diagnosed high-risk prostate cancer shows that about one-third of the patients present with advanced disease with lymph node or bone metastases. High specificity (96.5%) but low sensitivity (30.6%) was found for the diagnosis of pelvic lymph node metastasis. It has also recently been shown in a well-designed randomized prospective trial that 68Ga-PSMA-PET/CT had a 27% greater accuracy than conventional imaging with CECT and BS. High accuracy is also supported by the results from a recent retrospective study of the favorable 18F-PSMA-1007-PET/CT, which showed sensitivity for lymph node metastasis of 85.9% and a specificity of 99.5% in a setting of patients with predominantly primary PCa. So, when would it be time to implement PSMA-PET/CT for staging patients with primary PCa? The European guidelines report that it could be tempting to replace BS and CECT by more accurate tests such as PSMA-PET/CT in patients undergoing initial PCa staging. They are concerned, however, that the clinical benefit of detecting metastases at an earlier time-point is undetermined. Therefore, it is argued that results from randomized controlled trials evaluating the management and outcome of patients by state-of-the-art diagnostic methods should be awaited before a decision can be made to treat patients based on the results of these tests. However, the investigators are not aware of any other current studies running or being planned to evaluate the impact of replacing traditional imaging with up-to-date PSMA-PET/CT on patient outcomes such as survival and quality-of-life.

Aims and objectives

The overall aim of this project is to analyze the impact on survival and quality of life of using PSMA-PET/CT for PCa primary staging compared with conventional imaging. In a randomized design the investigators will compare 18F-PSMA-1007 PET/CT (interventional imaging) with CECT and NaF-PET/CT (conventional imaging) as regards progression-free survival and quality of life. In subgroup analyses, the investigators aim to analyze the accuracy of 18F-PSMA-PET/CT compared with conventional imaging and the added value of 18F-PSMA-PET/MRi for local staging.

Treatment strategies will be planned and registered in multidisciplinary team conferences based on the results of the scans and according to current guidelines. The strategies will be categorized into radical prostatectomy, curatively intended radiotherapy, palliative radiotherapy, androgen deprivation therapy, chemotherapy, and metastases-directed therapy. These treatment options can be used separately or combined.

QoL changes will be considered clinically relevant for an 8-point decline in global Functional Assessment of Cancer Therapy - Prostate (FACT-P). Other QoL analyses include the group difference in repeated measurement analyses, making use of data collected at baselinie and 2 time points the first year after diagnoses and later at specific time points, and these will be conducted using the European Quality of life - 5 Dimensions - 5 Levels (EQ-5D-5L) and Expanded Prostate Cancer Index Composite-26 (EPIC-26) (internationally accepted and validated questionnaires translated into danish).

ELIGIBILITY:
Inclusion Criteria:

* Has given informed consent to participate
* Can read and understand provided patient information material in Danish
* Biopsy verified PCa
* Any, some, or all of the following features:

  * Prostatic Specific Antigen (PSA) ≥ 20 ng/ml OR
  * Gleason Score ≥ 4+3 OR
  * Tumor stage clinically judged T2c cancer (cT2c) or above as determined by digital rectal exploration and/or transrectal ultrasonography
  * Suspicion of metastases clinically based on other findings
* Prostatic Specific Antigen (PSA) ≤ 200 ng/ml
* Staging by imaging warranted

Exclusion Criteria:

* Consent not given
* Inability to read and/or understand provided patient information in Danish
* Previously given consent but withdrawn for any reason
* Staging by imaging not warranted as judged clinically
* Allergy towards contents in the tracer solution

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (Group A vs. B) | 1 to 3 years after staging
  Time from treatment with curative intent to progression, eg. time from staging/curative treatment to PSA-value (or other clinical findings) deeming relapse.

SECONDARY OUTCOMES:
Treatment Strategy (Group A vs. B) | Immediately after staging - 1-2 months after the scan.
  Treatment strategy compared between the two groups. Rate of patients offered prostatectomy, curative radiotherapy, curative intended treatment, castration, up-front chemotherapy) in each group.
Quality of life according to questionnaires (Group A vs. B) | 1 to 3 years after staging. Questionnaire: Functional Assessment of Cancer Therapy - Prostate Cancer (FACT-P v. 4)
  Difference in quality of life between the two groups judged by patient reported outcomes in questionnaires, an 8 point difference is considered clinically relevant in FACT-P. Minimum 0 points and maximum 156 points for FACT-P, higher score is worse. Level of significance will be 5%.

OTHER OUTCOMES:
Accuracy NaF-PET/CT compared to PSMA-PET/CT for detection of metastases | Immediately after staging/up to 1 month after the scan.
  Difference in metastases detection between the two groups
Value of PSMA/MR for tumor staging and detection of lymph node and bone metastases in the pelvis. | After prostatectomy, up to 3 months after the scan.
  Comparing pathology results with PSMA-PET/MRi for evaluating tumor extension in the prostate gland, and lymph node and bone metastases in the pelvis.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Department of Radiology and Nuclear Medicine, Esbjerg
  - Department of Nuclear Medicine, Odense
  - Department of Nuclear Medicine, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Parker CC, James ND, Brawley CD, Clarke NW, Hoyle AP, Ali A, Ritchie AWS, Attard G, Chowdhury S, Cross W, Dearnaley DP, Gillessen S, Gilson C, Jones RJ, Langley RE, Malik ZI, Mason MD, Matheson D, Millman R, Russell JM, Thalmann GN, Amos CL, Alonzi R, Bahl A, Birtle A, Din O, Douis H, Eswar C, Gale J, Gannon MR, Jonnada S, Khaksar S, Lester JF, O'Sullivan JM, Parikh OA, Pedley ID, Pudney DM, Sheehan DJ, Srihari NN, Tran ATH, Parmar MKB, Sydes MR; Systemic Therapy for Advanced or Metastatic Prostate cancer: Evaluation of Drug Efficacy (STAMPEDE) investigators. Radiotherapy to the primary tumour for newly diagnosed, metastatic prostate cancer (STAMPEDE): a randomised controlled phase 3 trial. Lancet. 2018 Dec 1;392(10162):2353-2366. doi: 10.1016/S0140-6736(18)32486-3. Epub 2018 Oct 21. PMID 30355464
- [Background] Connor MJ, Smith A, Miah S, Shah TT, Winkler M, Khoo V, Ahmed HU. Targeting Oligometastasis with Stereotactic Ablative Radiation Therapy or Surgery in Metastatic Hormone-sensitive Prostate Cancer: A Systematic Review of Prospective Clinical Trials. Eur Urol Oncol. 2020 Oct;3(5):582-593. doi: 10.1016/j.euo.2020.07.004. Epub 2020 Sep 3. PMID 32891600
- [Background] Shen G, Deng H, Hu S, Jia Z. Comparison of choline-PET/CT, MRI, SPECT, and bone scintigraphy in the diagnosis of bone metastases in patients with prostate cancer: a meta-analysis. Skeletal Radiol. 2014 Nov;43(11):1503-13. doi: 10.1007/s00256-014-1903-9. Epub 2014 May 20. PMID 24841276
- [Background] Zacho HD, Jochumsen MR, Langkilde NC, Mortensen JC, Haarmark C, Hendel HW, Jensen JB, Petersen LJ. No Added Value of 18F-Sodium Fluoride PET/CT for the Detection of Bone Metastases in Patients with Newly Diagnosed Prostate Cancer with Normal Bone Scintigraphy. J Nucl Med. 2019 Dec;60(12):1713-1716. doi: 10.2967/jnumed.119.229062. Epub 2019 May 30. PMID 31147402
- [Background] Klingenberg S, Jochumsen MR, Ulhoi BP, Fredsoe J, Sorensen KD, Borre M, Bouchelouche K. 68Ga-PSMA PET/CT for Primary Lymph Node and Distant Metastasis NM Staging of High-Risk Prostate Cancer. J Nucl Med. 2021 Feb;62(2):214-220. doi: 10.2967/jnumed.120.245605. Epub 2020 May 22. PMID 32444374
- [Background] Hofman MS, Lawrentschuk N, Francis RJ, Tang C, Vela I, Thomas P, Rutherford N, Martin JM, Frydenberg M, Shakher R, Wong LM, Taubman K, Ting Lee S, Hsiao E, Roach P, Nottage M, Kirkwood I, Hayne D, Link E, Marusic P, Matera A, Herschtal A, Iravani A, Hicks RJ, Williams S, Murphy DG; proPSMA Study Group Collaborators. Prostate-specific membrane antigen PET-CT in patients with high-risk prostate cancer before curative-intent surgery or radiotherapy (proPSMA): a prospective, randomised, multicentre study. Lancet. 2020 Apr 11;395(10231):1208-1216. doi: 10.1016/S0140-6736(20)30314-7. Epub 2020 Mar 22. PMID 32209449
- [Background] Sprute K, Kramer V, Koerber SA, Meneses M, Fernandez R, Soza-Ried C, Eiber M, Weber WA, Rauscher I, Rahbar K, Schaefers M, Watabe T, Uemura M, Naka S, Nonomura N, Hatazawa J, Schwab C, Schutz V, Hohenfellner M, Holland-Letz T, Debus J, Kratochwil C, Amaral H, Choyke PL, Haberkorn U, Sandoval C, Giesel FL. Diagnostic Accuracy of 18F-PSMA-1007 PET/CT Imaging for Lymph Node Staging of Prostate Carcinoma in Primary and Biochemical Recurrence. J Nucl Med. 2021 Feb;62(2):208-213. doi: 10.2967/jnumed.120.246363. Epub 2020 Aug 17. PMID 32817141
- See also: NORDCAN: Cancer Incidence, Mortality, Prevalence and Survival, accessed 2018/09/09 — http://www.ancr.nu
- See also: Guidelines in Prostate Cancer — http://uroweb.org/guideline/prostate-cancer/
- See also: Danish clinical Guidelines for Prostate Cancer — http://ducg.dk/daproca-prostatacancer/kliniske-retningslinjer/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT05123300/Prot_SAP_000.pdf